CLINICAL TRIAL: NCT01353807
Title: Impact of Fish Oil Supplementation in 3rd Trimester of Pregnancy on Maternal and Offspring Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Fetal Programming, Denmark (Other)
Collaborators: National Institutes of Health (NIH) (NIH); The Danish Council for Strategic Research (Other); Danish Council for Independent Research (Other); Lundbech Foundation (Unknown); EU Commision, DG12 (Unknown)
Responsible Party: Sjurdur Frodi Olsen, Statens Serum Institut, Copenhagen, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: M-AA-20060182; R21AT004603 (NIH)
Record Dates: First submitted 2011-04-29; First posted 2011-05-16 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Preterm Delivery; Atopy; Metabolic Syndrome
Keywords: Fish oil; Pregnancy; RCT; Birth weight; Gestational age; Asthma and allergies; Metabolic syndrome; Obesity
MeSH Terms: conditions — Premature Birth; Metabolic Syndrome; Birth Weight; Asthma; Hypersensitivity; Obesity | interventions — Fish Oils; Pikasol; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fish oil supplementation (Active Comparator): These women received 4 1-g capsules of fish oil per day providing 2,7 grams long chain n-3 fatty acids per day, from gestation week 30 until delivery
  Interventions: Dietary Supplement: Fish oil
- Olive oil (Placebo Comparator): These women received 4 1-g capsules with olive oil per day from gestational week 30 until delivery
  Interventions: Dietary Supplement: Olive oil
- No oil supplement (No Intervention): These women received no capsules with oil

INTERVENTIONS:
Dietary Supplement: Fish oil — 4 1-g gelatine capsules per day providing 2,7 grams long chain n-3 fatty acids
  Other Names: Pikasol
  Arms: Fish oil supplementation
Dietary Supplement: Olive oil — 4 1-g gelatine capsules with virgin olive oil
  Arms: Olive oil

SUMMARY:
The aim of the trial is to investigate the effect of daily supplementation with 2.7 grams of long chain n-3 fatty acids during the third trimester of pregnancy. In 1990, 533 pregnant women, while they were in gestational week 30, were randomized to fish oil supplements providing the mentioned amount of long chain n-3 fatty acids, olive oil supplements, or no supplements; they were asked to take the supplements until delivery. Health outcomes were assessed during pregnancy and delivery. Further, offspring health and development has been examined during the ensuring two decades by making linkages to the rich Danish health and administrative registries, by asking the offspring to complete web-based questionnaires, and by examining the offspring physically.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women in gestation week 30

Exclusion Criteria:

* Bleeding episodes during pregnancy

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 533 (Actual)
Dates: Start 1989-11; Primary Completion 1990-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Gestation length | 1989-1990 (1 year)
  We assesed impact of fish oil supplementation in pregnancy on timing of spontaneous delivery

CONTACTS AND LOCATIONS:
Overall Officials: Sjurdur F. Olsen, MD, Principal Investigator — Statens Serum Institut
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Result] Olsen SF, Sorensen JD, Secher NJ, Hedegaard M, Henriksen TB, Hansen HS, Grant A. Randomised controlled trial of effect of fish-oil supplementation on pregnancy duration. Lancet. 1992 Apr 25;339(8800):1003-7. doi: 10.1016/0140-6736(92)90533-9. PMID 1349049
- [Result] Olsen SF, Osterdal ML, Salvig JD, Mortensen LM, Rytter D, Secher NJ, Henriksen TB. Fish oil intake compared with olive oil intake in late pregnancy and asthma in the offspring: 16 y of registry-based follow-up from a randomized controlled trial. Am J Clin Nutr. 2008 Jul;88(1):167-75. doi: 10.1093/ajcn/88.1.167. PMID 18614738
- [Result] Rytter D, Bech BH, Christensen JH, Schmidt EB, Henriksen TB, Olsen SF. Intake of fish oil during pregnancy and adiposity in 19-y-old offspring: follow-up on a randomized controlled trial. Am J Clin Nutr. 2011 Sep;94(3):701-8. doi: 10.3945/ajcn.111.014969. Epub 2011 Jul 20. PMID 21775563
- [Result] Rytter D, Schmidt EB, Bech BH, Christensen JH, Henriksen TB, Olsen SF. Fish oil supplementation during late pregnancy does not influence plasma lipids or lipoprotein levels in young adult offspring. Lipids. 2011 Dec;46(12):1091-9. doi: 10.1007/s11745-011-3606-5. Epub 2011 Aug 27. PMID 21874272
- [Result] Rytter D, Christensen JH, Bech BH, Schmidt EB, Henriksen TB, Olsen SF. The effect of maternal fish oil supplementation during the last trimester of pregnancy on blood pressure, heart rate and heart rate variability in the 19-year-old offspring. Br J Nutr. 2012 Oct 28;108(8):1475-83. doi: 10.1017/S0007114511006799. Epub 2012 Feb 7. PMID 22313729
- See also: Protocol and correspondences — http://cfp-research.com/Research/Publications/Sjurdur%20F%20Olsen.aspx